CLINICAL TRIAL: NCT07285772
Title: Clinical Performance of Various Bilayer Biomimetic Resin Composite Strategies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Abd El Ghany Mohammed, Doctor, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: biomimetic resin composite
Record Dates: First submitted 2025-11-22; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Composite Restoration; Composites Resins
Keywords: Clinical; Biomimetic; Composite; Class I
MeSH Terms: interventions — flowable hybrid composite

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- EverX Posterior composite (Experimental): Short fiber-reinforced composite
  Interventions: Other: short fiber reinforced composite , long fiber reinforced composite, light cure glass, flowable composite
- Ribbond (Experimental): Long fiber-reinforced composite
  Interventions: Other: short fiber reinforced composite , long fiber reinforced composite, light cure glass, flowable composite
- Riva SDI (Experimental): glass ionomer restorative material
  Interventions: Other: short fiber reinforced composite , long fiber reinforced composite, light cure glass, flowable composite
- G-aenial universal Flo (Experimental): flowable composite
  Interventions: Other: short fiber reinforced composite , long fiber reinforced composite, light cure glass, flowable composite

INTERVENTIONS:
Other: short fiber reinforced composite , long fiber reinforced composite, light cure glass, flowable composite — All patients received four various bilayer biomimetic restorations in four groups (n = 40) as follows: Group I: short fiber reinforced composite (everX Posterior); ); Group II: long fiber reinforced composite (Ribbond Inc., USA); Group III: glass ionomer restorative materials (Riva SDI); and Group IV: flowable composite (G-aenial universal).

SUMMARY:
The purpose of this study was to evaluate several bilayer biomimetic composite resin techniques in class I cavities over the course of 18 months in a randomized, double-blind clinical trial.

DETAILED DESCRIPTION:
To make resin composite restorations more resistant to cracking in cavities that are under a lot of stress, some have proposed using fiber reinforcement. This proposal is supported by numerous prior investigations that have demonstrated the efficacy of these repairs. By adjusting their orientation, fibers can control the pressures brought on by polymerization shrinkage. Therefore, marginal microleakage has been reduced in comparison to conventional resin composites. One way the material's fibers improve its structural characteristics is by preventing cracks from propagating. Composites are ideal for direct restorations of large cavities in healthy teeth and teeth that have had endodontic treatment because the fiber structure improves their mechanical properties. Moreover, in 2021, a comprehensive analysis of research found that resin composite restorations reinforced with fibers had better adaptability and higher fracture resistance than the standard ones.

ELIGIBILITY:
Inclusion Criteria:

* Proper oral hygiene
* Availability for follow-up periods

Exclusion Criteria:

* Endodontically treated or non-vital teeth
* Parafunctional habits such as tooth clenching or grinding

Ages: 35 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-10-10 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
The primary outcomes are: surface luster, marginal staining, marginal adaptation, fracture, secondary caries, and postoperative sensitivity. | 18 months
  Clinical assessment was carried out according to the World Dental Federation (FDI) by two calibrated evaluators at baseline and at 6, 9, 12, and 18 months. All of the restorations were ranked according to how well they met the criteria: clinically excellent or very satisfactory, clinically satisfactory, clinically satisfactory, or clinically inadequate. Clinical success was defined as a score of 1, 2, or 3, and failure was indicated by scores of 4 or 5. A powerful light source was used to conduct the visual inspection of the parameters. A magnifying dental loupe was utilized for this purpose. The Friedman test was conducted to evaluate intragroup comparisons of the same restoration outcomes through different follow-up periods. The Kruskal-Wallis test was utilized to assess intergroup comparisons between different restorations during the same follow-up period.

CONTACTS AND LOCATIONS:
Locations (1):
- Restorative Department, Faculty of Dentistry, Tanta University, Tanta, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tanner J, Tolvanen M, Garoushi S, Sailynoja E. Clinical Evaluation of Fiber-Reinforced Composite Restorations in Posterior Teeth - Results of 2.5 Year Follow-up. Open Dent J. 2018 Jun 29;12:476-485. doi: 10.2174/1874210601812010476. eCollection 2018. PMID 30069257
- [Background] ElAziz RH, Mohammed MM, Gomaa HA. Clinical Performance of Short-fiber-reinforced Resin Composite Restorations vs Resin Composite Onlay Restorations in Complex Cavities of Molars (Randomized Clinical Trial). J Contemp Dent Pract. 2020 Mar 1;21(3):296-303. PMID 32434978
- [Background] Metwaly AA, Elzoghby AF, Abd ElAziz RH. Clinical performance of polyethylenefiber reinforced resin composite restorations in endodontically treated teeth: (a randomized controlled clinical trial). BMC Oral Health. 2024 Oct 24;24(1):1285. doi: 10.1186/s12903-024-05009-8. PMID 39448991
- [Background] Mohamed MH, Abouauf EA, Mosallam RS. Clinical performance of class II MOD fiber reinforced resin composite restorations: an 18-month randomized controlled clinical trial. BMC Oral Health. 2025 Jan 30;25(1):159. doi: 10.1186/s12903-025-05521-5. PMID 39881262